CLINICAL TRIAL: NCT06647849
Title: Interest of Simulation Training on the Announcement of Early Pregnancy Loss on the Psychological Impact of the Patients
Acronym: MISC-TRAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 49RC21_0257; 2024-A01244-43 (Other: Agence nationale de sécurité du médicament et des produits de santé)
Record Dates: First submitted 2024-10-09; First posted 2024-10-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-06

CONDITIONS: Early Pregnancy Loss; Spontaneous Miscarriage
Keywords: spontaneous miscarriage; early pregnancy loss; training for interns
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Multicenter Studies as Topic

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study will be single-blind. The patient will not know the intern's level of training (trained or untrained).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm "with training" (Experimental): Arm "with training": centers whose interns receive simulation training in the announcement of early spontaneous miscarriage between the 2 inclusion phases.
  Interventions: Procedure: centers whose interns receive simulation training in the announcement of early spontaneous miscarriage between the 2 inclusion phases
- "Untrained" arm (Other): "Untrained" arm: centers with standard in-house management of spontaneous miscarriage/pregnancy arrested in the emergency department.
  Interventions: Other: centers with standard in-house management of spontaneous miscarriage/pregnancy arrested in the emergency department

INTERVENTIONS:
Procedure: centers whose interns receive simulation training in the announcement of early spontaneous miscarriage between the 2 inclusion phases — The simulation training sessions for the announcement consultation are set up directly in the centers participating in the "with training" arm of the study, after the first phase of patient inclusion. These sessions will take place "in situ" in the center's maternity ward, and will be run by a single team trained in simulation and announcement.
  This team of trainers is identical for all centers randomized in the "with training" arm, and is made up of two trainers: an obstetrician-gynecologist and a psychologist.
  Arms: Arm "with training"
Other: centers with standard in-house management of spontaneous miscarriage/pregnancy arrested in the emergency department — In the participating centers included in the "no training" arm, interns will have no specific training in announcement. Patients will receive information concerning the diagnosis of a terminated pregnancy or miscarriage from interns not trained in simulation.
  During the course of the study, training in the announcement of a miscarriage will be offered to interns from centers in the "no training" group.
  Arms: "Untrained" arm

SUMMARY:
Early pregnancy loss (or spontaneous miscarriage) is the loss of a pregnancy before 14 weeks of amenorrhea. Its incidence is estimated at between 10 and 15%, and increases with maternal age.

Early pregnancy loss can have major psychological consequences for the woman, her partner and the couple in the aftermath, as well as on the experience and progress of a future pregnancy.

In France, the vast majority of miscarriages are diagnosed in gynecological emergencies by interns still in training. Interns, sometimes at the beginning of their training, may find it difficult to announce a miscarriage, and may do so in a way that is clumsy or not adapted to the woman's emotions, which can lead to a bad experience for her. This bad experience could lead to psychological distress, post-traumatic stress and/or impair future fertility.

The initiators of this project have already carried out a before-and-after, single-center study, showing a significant improvement in the specific Perinatal Grief Scale score following specific training for interns in first-trimester pregnancy loss.

To date, no multicenter randomized study has been conducted to assess the impact of first-trimester pregnancy loss on women's psychological experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient presenting to gynaecological emergency department
* Patient with a diagnosis of terminated pregnancy or spontaneous expulsion of a pregnancy < 14 weeks' amenorrhea
* Patient whose spontaneous miscarriage was announced by an intern
* Patient affiliated to or benefiting from a social security scheme
* Patient having signed an informed consent form

Exclusion Criteria:

* Unwanted pregnancy
* Spontaneous hemorrhagic miscarriage requiring surgical management
* Ectopic pregnancy
* Miscarriage resulting from assisted reproduction treatment
* Patient with history of miscarriage ≥ 3
* Poor understanding of the French language
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person subject to a legal protection measure
* Person unable to give consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-05-11 (Estimated); Study Completion 2027-06-11 (Estimated)

PRIMARY OUTCOMES:
evaluate the impact of specific training for interns in simulated early miscarriage announcements on patients' psychological experiences | The primary endpoint was the significant change in the Perinatal Grief Scale at 3 months post-miscarriage linked to the implementation of the simulation training

SECONDARY OUTCOMES:
Evaluation of the impact on the psychological experience of short-term miscarriage at 1 month | Modification of the "Impact of event scale-revised" post-traumatic stress score at 1 month
evaluation of the patient's feelings about the miscarriage announcement made by the intern at 1 month | Modification of the patient's perception of the announcement of the miscarriage by the resident, using a 1-month questionnaire
Assessing the impact of long-term miscarriage on psychological experience | Modification in the Perinatal Grief Scale score at 6 and 12 months post-miscarriage linked to the introduction of simulated announcement training
Fertility assessment at 6 and 12 months | Time to decision to have a new pregnancy and increase in clinical pregnancy rates, progressive pregnancy rates > 14 weeks' amenorrhea at 6 and 12 months
Comparing the difference of " Impact of event scale-revised" score in patients depending on whether they are cared for by an intern whose most recent training in prognosis was less than or more than 6 months ago | 18 months
Comparing the difference of " Impact of event scale-revised" score in patients depending on whether they were cared for by an intern who had received a single training course less than 6 months old, or by an intern who had received two training courses | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Legendre, MD, PhD, Study Director — University Hospital of Angers
Locations (28):
- France (28):
  - University Hospital of Amiens, Amiens
  - University Hospital of Angers, Angers
  - University Hospital of Bordeaux, Bordeaux
  - University Hospital of Brest, Brest
  - Femme Mere Enfant Hospital, Bron
  - University Hospital of Caen, Caen
  - CH Chalon-sur-Saône, Chalon-sur-Saône
  - CH Cholet, Cholet
  - University Hospital of Clermont-Ferrand, Clermont-Ferrand
  - University Hospital of Dijon, Dijon
  - CHU Grenoble, Grenoble
  - Vendée Departmental Hospital center, La Roche-sur-Yon
  - Le Mans Hospital, Le Mans
  - Jeanne de Flandre Hospital, Lille
  - University Hospital of Limoges, Limoges
  - Hopital Nord (Marseille Public University Hospital System), Marseille
  - La Conception Hospital (Marseille Public University Hospital System), Marseille
  - University Hospital of Montpellier, Montpellier
  - University Hospital of Nancy, Nancy
  - University Hospital of Nantes, Nantes
  - CHU Nice, Nice
  - University Hospital of Nimes, Nîmes
  - CHU Orléans, Orléans
  - Poissy intercommunal hospital center, Poissy
  - University Hsopital of Reims, Reims
  - University Hospital of Rennes, Rennes
  - University Hospital of Rouen, Rouen
  - University Hospital of Saint Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No